CLINICAL TRIAL: NCT02280837
Title: An Observational Study to Examine the Relationship Between GLP-1 Insufficiency and Severity of Coronary Artery Disease in Patients Enrolled in BOREAS Registry, a Prospective Registry of Cardiovascular and Renal Diseases. : Is GLP-1 Insufficiency a Residual Risk in Coronary Artery Disease?
Brief Title: Is Glucagon-like Peptide-1 Insufficiency a Residual Risk in Coronary Artery Disease?
Status: Completed | Type: Observational
Sponsor: Sapporo Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 262-83
Record Dates: First submitted 2014-10-26; First posted 2014-11-03 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease
Keywords: GLP-1
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with suspected or diagnosed coronary artery disease
  Interventions: Other: Determination of plasma GLP-1 level

INTERVENTIONS:
Other: Determination of plasma GLP-1 level — Determination of GLP-1 level in samples of oral glucose tolerance tests

SUMMARY:
In this study, the investigators hypothesized that significant proportion of patients with coronary artery disease (CAD) has reduced capacity of glucagon-like peptide-1 (GLP-1) secretion, which is detectable as blunted response of plasma active GLP-1 level to oral glucose loading and that reduced GLP-1 secretory function is associated with increased severity of coronary artery stenosis but not with classic risk factors for CAD. To test this hypothesis, the investigators will analyze correlation between GLP-1 secretory capacity and severity of coronary artery stenosis determined by Gensini Score (GS), an established score system for coronary artery stenoses. Additionally, the investigators will analyze relationship between level of "total" GLP-1 and severity of coronary artery stenosis to determine how it is different from the active GLP-1 - coronary stenosis relationship.

DETAILED DESCRIPTION:
Recently, the investigators found that a significant proportion of subjects in a general population shows attenuated secretion of active GLP-1 in response to oral glucose loading and that the insufficient secretion of GLP-1 was independently associated with elevation of blood pressure (BP) (Yoshihara et al. PLoS One 2013;8:e67578). In that study, it was also found that the amount of GLP-1 secreted after glucose loading was not correlated with any of conventional serum lipid parameters (i.e., triglyceride, LDL-cholesterol and HDL-cholesterol) or plasma insulin level. These findings suggest that insufficiency of GLP-1 secretion may promote atherosclerosis and formation of coronary plaques. Furthermore, lack of correlation between response of active GLP-1 secretion and serum lipids or plasma insulin indicates that insufficient secretion of active GLP-1 may be a hidden risk factor of atherosclerotic vascular disease. Based on those results in a previous study, the investigators designed the present study.

The present study is a single-centered (Sapporo Medical University Hospital), observational study enrolling patients who will be admitted to our institute for coronary angiogram. Written informed consent will be obtained from patients on admission. Patients will receive demographic measurements, blood sampling for routine serum biochemistry and detailed analyses of serum lipids (such as apolipoproteins, remnant-like lipoprotein particle and oxidized-LDL-cholesterol) after overnight fast and oral glucose tolerance test (OGTT). In OGTT, blood will be sampled for assay of glucose, insulin, active GLP-1 and total GLP-1 before, 30 min, 60 min, and 120 min after oral 75 g-glucose loading. Capacity of GLP-1 secretion will be determined as area under the curve of plasma GLP-1 level (AUC-GLP-1). All study subjects will undergo coronary angiogram and severity of coronary artery stenosis will be quantified by Gensini score (GS). Relationship between GS, AUC-active-GLP-1 or AUC-total-GLP-1, blood pressure, serum lipid parameters, and indices of insulin resistance (homeostasis model assessment as an index of insulin resistance and Matsuda-Defronzo index) will be examined by use of univariate and multivariate regression analyses to determine whether AUC-active-GLP-1 or AUC-total-GLP-1 is an independent determinant of coronary artery stenosis. This study will be conducted as one of projects in BOREAS registry, a non-interventional, multicenter registry of cardiovascular and/or renal diseases conducted by our institute and affiliated hospitals.

The time frame for which the outcome measures is assessed: Informed consent on Hospital day 1, Demographic examinations and blood and urine tests on Hospital day 1 and day 2, OGTT on Hospital day 2 or day 3, Coronary angiogram and scoring coronary stenoses on Hospital day 3 or a later day within 14 days after admission (patients who could not undergo angiogram within 14 days after admission by incidental causes will be excluded), Acquisition of data necessary for analyses on Day 9-17 (Data set of each patients, including remnant-like protein particle, ApoA1, ApoB, and ApoE, will be mostly completed within approximately 9-17 days after admission. Samples for determination of GLP-1 will be stored at -80 C until assay).

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic patients (HbA1c <6.5%) with suspected or diagnosed CAD at ages of 35-80 years who are hospitalized for coronary angiogram will included in this study. - No change in medications (if any) for dyslipidemia within 3 month prior to admission is also a criterion for inclusion.

Exclusion Criteria:

* Diabetic patients whose HbA1c is higher than 6.5% or who have received insulin or hypoglycemic agents and those who need immediate pharmacological treatments after admission will be excluded.
* Patients with history of PCI also will be excluded.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-diabetic patients with suspected or diagnosed CAD who are hospitalized for coronary angiogram will be enrolled in this study. The patients are expected to be similar to those who have visited our institute recently; approximately 28% of patients with CAD are diabetics, and one third of them are medically untreated at the time of their first visit. In recent years, 500-600 patients have undergone coronary angiography per year in this institute, and approximately 50% of them were without history of percutaneous coronary interventions (PCI) or coronary bypass surgery. Hence, approximately 180-210 patients per year will be candidates for the present project.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Severity of coronary artery stenosis expressed as Gensini Score determined by coronary angiography | at the time of coronary angiogram: Coronary angiogram will be performed on Hospital day 3 or a later day within 14 days after admission.

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuji Miura, MD, PhD, Principal Investigator — Sapporo Medical University
Locations (1):
- Sapporo Medical University, School of Medicine, Sapporo, Hokkaido, Japan